CLINICAL TRIAL: NCT00060632
Title: A Phase I, Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability, and Maximum Tolerated Dose of Weekly Administration of AP23573, an mTOR Inhibitor, in Patients With Refractory or Advanced Malignancies
Brief Title: Safety Study of Ridaforolimus in Patients With Advanced, Refractory or Recurrent Malignancies (MK-8669-001 AM5)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-001; AP23573-02-101
Record Dates: First submitted 2003-05-08; First posted 2003-05-12 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Tumors; Lymphoma; Multiple Myeloma
Keywords: Advanced, refractory or recurrent solid tumors
MeSH Terms: conditions — Neoplasms; Lymphoma; Multiple Myeloma | interventions — ridaforolimus

ARMS (6):
- Cohort 1: Ridaforolimus 6.25 mg (Experimental)
  Interventions: Drug: ridaforolimus
- Cohort 2: Ridaforolimus 12.5 mg (Experimental)
  Interventions: Drug: ridaforolimus
- Cohort 3: Ridaforolimus 25 mg (Experimental)
  Interventions: Drug: ridaforolimus
- Cohort 4: Ridaforolimus 50 mg (Experimental)
  Interventions: Drug: ridaforolimus
- Cohort 5: Ridaforolimus 100 mg (Experimental)
  Interventions: Drug: ridaforolimus
- Cohort 6: Ridaforolimus 75 mg (Experimental)
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — Administered intravenously once weekly for 4 weeks (1 cycle).
  In the absence of disease progression or unacceptable toxicity, patients could continue to receive additional cycles.
  Other Names: AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
Phase 1 trial to determine the safety, tolerability and maximum tolerated dose (MTD) of ridaforolimus in patients with refractory or recurrent malignancies, including myeloma and lymphoma.

DETAILED DESCRIPTION:
The primary objectives of the study are to determine the safety, tolerability, and MTD of ridaforolimus when administered once weekly for 4 weeks (4 week cycle). The secondary objectives of the study are to characterize the pharmacokinetic profile of ridaforolimus, to evaluate potential pharmacodynamic markers of ridaforolimus, and to obtain preliminary information on the antineoplastic activity of ridaforolimus.

Protocol Outline: This is a dose-escalation study. Patients receive ridaforolimus over 30 minutes by intravenous infusion once weekly for 8 weeks (two 4-week cycles). If tolerated, a total of at least 2 cycles will be administered (8-week treatment period). Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

(Patients must meet each of the following criteria to be eligible for participation in the study).

* Male or female patients, ≥ 18 years of age.
* Patients with a documented measurable or evaluable malignancy, including myeloma or lymphoma, that is recurrent, advanced, or metastatic.
* Patients with disease that is currently refractory to, or not amenable to, standard therapy.
* Patients with disease that is currently not amenable to surgical intervention.
* Patients with Karnofsky performance status of ≥ 70% (Eastern Cooperative Oncology Group [ECOG] performance status of 0 or 1) and an anticipated life expectancy of ≥ 3 months.
* Patients either not of childbearing potential, or agreeing to use a medically effective method of contraception.
* Patients with the ability to understand and give written informed consent.

Exclusion Criteria:

(Patients meeting any of the following criteria are ineligible for participation in the study)

* Women who are pregnant or lactating.
* Patients with primary central nervous system (CNS) malignancies. Patients with leukemia, any form.
* Patients with certain hematologic abnormalities.
* Patients with certain serum chemistry abnormalities at baseline.
* Patients with known or suspected hypersensitivity to either drugs formulated with polysorbate 80 (Tween 80) or any other excipient contained in the test drug formulation.
* Patients with known hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin).
* Patients with significant cardiovascular disease.
* Patients with active CNS metastases (or leptomeningeal disease) not controlled by prior surgery or radiotherapy. Note: Patients with treated brain metastases will be eligible if they are on a stable dose of corticosteroids or are without change in brain disease status for at least 4 weeks following related therapy (e.g., whole brain radiation, surgery).
* Patients with known human immunodeficiency virus (HIV) infection.
* Patients with any active infection.
* Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 2 weeks prior to study entry. Note: Patients having undergone recent placement of a central venous access port will be considered eligible for enrollment if they have recovered.
* Patients who have any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the test drug.
* Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies.
* Patients with the inability, in the opinion of the Investigator, to comply with the protocol requirements.

Drugs and Other Treatments to be Excluded (Either during or within 4 weeks prior to study entry, unless otherwise noted)

* Chemotherapeutic agents (standard or experimental).
* Other antineoplastic agents.
* Immunotherapy (including vaccines) or biological response modifier therapy.
* Systemic replacement hormonal therapy for life-threatening non-oncology diseases.
* Herbal preparations or related over-the-counter (OTC) preparations containing herbal ingredients (e.g., St John's Wort) during or within 2 weeks prior to study entry.
* Any prior therapy with rapamycin, CCI-779, or any other rapamycin analog.
* Any other experimental therapy during the course of the study.
* Radiotherapy for the primary malignancy or metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Cycle 1 (within the first 4 weeks)
Number of Participants Reporting Adverse Events (AE) | Throughout study duration and up to approximately 1 month after the last dosing cycle (Cycle 1 Day 1 to approximately 10 months)
Number of Participants Discontinuing Due to AEs | Throughout study duration (Cycle 1 Day 1 to approximately 9 months)

SECONDARY OUTCOMES:
Best Overall Tumor Response | 8 weeks
Maximum Concentration (Cmax) of Ridaforolimus | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1
Area Under the Curve (AUC[0 to Infinity]) of Ridaforolimus | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1
Apparent Terminal Half-Life (t1/2) of Ridaforolimus | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1
Clearance (CL) of Ridaforolimus | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1
Volume of Distribution at Steady State (Vss) of Ridaforolimus | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1
Phosphorylated 4E Binding Protein 1 (Phospho-4E-BP1) Blood Levels | Screening, Cycle 1 Days 1, 2, 3, 6/7, 8; Cycle 2 Day 1

REFERENCES:
- [Background] Hartford CM, Desai AA, Janisch L, Karrison T, Rivera VM, Berk L, Loewy JW, Kindler H, Stadler WM, Knowles HL, Bedrosian C, Ratain MJ. A phase I trial to determine the safety, tolerability, and maximum tolerated dose of deforolimus in patients with advanced malignancies. Clin Cancer Res. 2009 Feb 15;15(4):1428-34. doi: 10.1158/1078-0432.CCR-08-2076. PMID 19228743